CLINICAL TRIAL: NCT01966172
Title: Multimodal Opiate-sparing Analgesia Versus Traditional Opiate Based Analgesia After Cardiac Surgery, a Randomized Controlled Trial
Brief Title: Multimodal Analgesic Treatment Versus Traditional Morphine Analgesia After Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Sulman Rafiq, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Smerte1
Record Dates: First submitted 2013-09-30; First posted 2013-10-21 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-10

CONDITIONS: Analgesia; Postoperative Pain
Keywords: NSAID, gabapentin, multimodal, morphine, dexamethasone, cardiac surgery, postoperative pain, analgesia.
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Ibuprofen; Gabapentin; Morphine; Acetaminophen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multimodal (Experimental): oral Ibuprofen 400mg 4 times daily oral Gabapentin 300mg twice daily oral Paracetamol 1000mg 4 times daily
  Interventions: Drug: Ibuprofen; Drug: Gabapentin; Drug: Paracetamol
- Morphine (Active Comparator): oral Morphine 10mg 4 times daily oral paracetamol 1000mg 4 times daily
  Interventions: Drug: Morphine; Drug: Paracetamol

INTERVENTIONS:
Drug: Ibuprofen — oral ibuprofen 400mg 4 times daily
  Other Names: non-selective Non-steroid antiinflammatory drug (NSAID)
  Arms: Multimodal
Drug: Gabapentin — Oral Gabapentin 300mg twice daily
  Arms: Multimodal
Drug: Morphine — 10 mg morphine orally 4 times daily
  Other Names: An opiod
  Arms: Morphine
Drug: Paracetamol — oral paracetamol 1000mg four times daily

SUMMARY:
To test if multimodal analgesia with different analgesic medication offer better pain relief, lesser side effects and is safe compared to conventionel opiod analgesia after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* age>18
* any cardiac procedure with sternotomy
* able to give informed consent

Exclusion Criteria:

* cardiac surgery without sternotomy
* peripheral neuropathy
* neurological disease
* psychiatric illness
* history of GI bleeding
* chronic pain (i.e. back pain, cancer, arthritis)
* serum creatinine >150 μmol/l
* hepatic disease with elevated liver enzymes (SGPT and SGOT elevated to 1.5 times maximum normal value)
* allergic to study medication
* alcohol abuse
* abuse of narcotics or medication
* pregnancy
* participation in other clinical trials
* insufficient language skills
* In addition intensive care unit (ICU) stay for more than 24 hours was used as a pre-defined post randomization exclusion criteria, because prolonged ICU stay and ventilator treatment would interfere with study analgesic protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-03; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of analgesic effect by 11-NRS scale | 4th postoperative day
  assessement of analgesic effect for the first 4 days after surgery

SECONDARY OUTCOMES:
Additional analgesic consumption | 4th postoperative day
Hospital stay in days. | days until discharge
Evaluation of side-effects by daily questionnaire | 4th postoperative day
Cardiac complications | 30th postoperative day
  i.e. Myocardial infarction(MI), postoperative pericardial effusion, heart failure requiring inotropic support , atrial fibrillation.
Other complications | 30th postoperative day
  i.e. cerebral (stroke, bleeding), GI(bleeding), blood component requirements and sternal complications.
30 day Mortality | 30th postoperative day
  Death from all causes.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Skov Olsen, MD,PhD,DMSc, Principal Investigator — Rigshospitalet, Denmark; Sulman Rafiq, MD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Rafiq S, Steinbruchel DA, Wanscher MJ, Andersen LW, Navne A, Lilleoer NB, Olsen PS. Multimodal analgesia versus traditional opiate based analgesia after cardiac surgery, a randomized controlled trial. J Cardiothorac Surg. 2014 Mar 20;9:52. doi: 10.1186/1749-8090-9-52. PMID 24650125